CLINICAL TRIAL: NCT00619424
Title: A Phase I Study of Pazopanib in Combination With Either Erlotinib or Pemetrexed in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study Of Pazopanib With Either Erlotinib Or Pemetrexed In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEG109607
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: erlotinib; pharmacokinetics; Solid tumors; pemetrexed; anti-angiogenesis; pazopanib (GW786034); cytokine and angiogenic factors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pazopanib; Erlotinib Hydrochloride; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pazopanib + erlotinib (Experimental): Pazopanib and erlotinib are to be combined at different specified dose levels until an optimally tolerated dose level is identified. Pazopanib, a multi-targeted tyrosine kinase inhibitor of VEGFR-1, -2, and -3, PDGFR-alpha and beta, and c-kit and erlotinib, an epidermal growth factor (EGFR) inhibitor, are to be combined in an effort to simultaneously block two tightly woven cell signaling pathways.
  Interventions: Drug: pazopanib; Drug: erlotinib
- pazopanib + pemetrexed (Experimental): Pazopanib and pemetrexed are to be combined at different specified dose levels until an optimally tolerated dose regimen is identified. Combination of an anti-VEGF therapy (such as bevacizumab) with systemic chemotherapy has demonstrated increased clinical efficacy in comparison with systemic chemotherapy alone in several malignancies. Hence, pazopanib, a multi-targeted tyrosine kinase inhibitor of VEGFR-1, -2, and -3, PDGFR-alpha and beta, and c-kit, was chosen to be combined with pemetrexed, a chemotherapeutic agent that inhibits the enzyme thymidylate synthase, in an effort to determine if an anti-angiogenesis inhibitor would enhance the activity of the approved chemotherapeutic agent pemetrexed.
  Interventions: Drug: pazopanib; Drug: pemetrexed

INTERVENTIONS:
Drug: pazopanib — Oral tablet administered daily in dosages of 400 - 800 mg.
Drug: erlotinib — oral tablet taken daily in dosages of 100-150 mg.
  Arms: pazopanib + erlotinib
Drug: pemetrexed — IV chemotherapeutic agent administered every 21 days in dosages of 400-500 mg/m2
  Arms: pazopanib + pemetrexed

SUMMARY:
This is an open-label, two-arm, Phase I, dose escalation study to evaluate the safety and tolerability and to determine the maximum tolerated dose (MTD) of pazopanib in combination with erlotinib (Arm A) or pazopanib in combination with pemetrexed (Arm B) in patients with advanced solid tumors. Patients will be enrolled in cohorts of 3 (in each arm) to receive escalating doses of pazopanib and erlotinib or pazopanib and pemetrexed. Dose escalation schemas for each study arm are described in the protocol. For each arm, the MTD regimen will be defined as the highest dose combination of the agents where no more than one out of six patients experiences a dose-limiting toxicity. Six to twelve additional patients in each arm will be studied with the MTD regimen to evaluate toxicity and pharmacokinetics. In arm A (erlotinib), a run-in phase with each drug separately will allow an evaluation of pharmacokinetics with each drug separately and also for the two drugs in combination. This will allow an assessment of potential drug-drug interactions. Pharmacokinetic endpoints will be AUC, Cmax, tmax and t1/2 of pazopanib, erlotinib, and pemetrexed, as well as pemetrexed clearance before and after administration of pazopanib in the extension cohort of Arm B. Antitumor activity will be assessed using RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

A subject will be considered eligible for inclusion in this study only if all of the following criteria are met:

* Subjects must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow up.

  ·Procedures conducted as a part of routine clinical management of the subject (e.g., blood count, imaging study) and obtained prior to signed informed consent may be utilized for Screening or Baseline purposes provided these tests are obtained as specified in the protocol.
* Histologically- or cytologically-confirmed diagnosis of advanced solid tumor that has failed standard therapy or for which there is no standard therapy. Subjects for whom erlotinib or pemetrexed are standard therapy may also be entered.
* Age ≥18 years.
* ECOG Performance status must be ≤1.
* Adequate organ system function as defined in Table 9. System (Laboratory Values)

Hematologic:

Absolute neutrophil count (ANC) ((≥1.5 X 10^9/L)) Hemoglobin (≥10 g/dL) Platelets (≥ 100 X 10^9/L) Prothrombin time (PT) or international normalized ration (INR) (≤ 1.2 X upper limit of normal (ULN)) Activated partial thromboplastin time (APTT) (≤ 1.2 X ULN)

Hepatic:

Total bilirubin (≤1.5 X ULN) AST and ALT (≤ 2.5 X ULN)

Renal:

Serum creatinine (≤ 1.5 mg/dL) Or, if greater than 1.5 mg/dL Calculated creatinine clearance (≤ 50 mL/min) Urine Protein to Creatinine Ratio (UPC)2 < 1

1. Subjects may not have had a transfusion within 7 days of screening assessment.
2. If UPC ≥ 1, then a 24-hour urine protein must be assessed and 24-hour urine protein must be <1 g protein to be eligible.

   * Measurable disease on CT scan.
   * A female subject is eligible to enter and participate in the study if she is of: • Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any woman who has had:• A hysterectomy
   * A bilateral oophorectomy (ovariectomy)
   * A bilateral tubal ligation
   * Is post-menopausal:
   * Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value >40mIU/mL and an estradiol value <40pg/mL (<140pmol/L).
   * Subjects must discontinue HRT prior to study enrollment due to the potential for inhibition of CYP enzymes that metabolize estrogens and progestins (see Section 8). For most forms of HRT, at least 2 4 weeks must elapse between the cessation of HRT and determination of menopausal status; length of this interval depends on the type and dosage of HRT. If a female subject is determined not to be post-menopausal, they must use adequate contraception, as defined immediately below.
   * OR of Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:
   * An intrauterine device with a documented failure rate of less than 1% per year.
   * Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
   * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product.
   * Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).

Note: Oral contraceptives are not reliable due to potential drug-drug interactions.

Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

A male with a female partner of childbearing potential is eligible to enter and participate in the study if he uses a barrier method of contraception or abstinence during the study.

* For Arm B (pemetrexed plus pazopanib) subjects:
* Must be able to permanently discontinue aspirin dose of ≥1.3 g/day for ≥10 days before through ≥10 days after pemetrexed disodium treatment. All subjects should be able to interrupt intake of NSAIDs with longer half lives (e.g., nabumetone, piroxicam, oxaprozin) for at least 5 days before, the day of, and 2 days following pemetrexed disodium administration.
* With mild to moderate renal insufficiency (CrCl from 50-79mL/min) should avoid taking NSAIDs with short elimination half lives (e.g., fenoprofen, indomethacin, ketoprofen, tolmetin, meclofenamate) for a period of 2 days before, the day of, and 2 days following administration of pemetrexed disodium.

Exclusion Criteria:

* Prior use of pazopanib, erlotinib (for subjects in Arm A), or pemetrexed (for subjects in Arm B).
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for one week prior to date of first dose of study drug. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required for all subjects.
* Clinically significant gastrointestinal abnormalities which might interfere with oral dosing, including but not limited to:
* Malabsorption syndrome
* Major resection of the stomach or small bowel that could affect the absorption of study drug
* Active peptic ulcer disease
* Inflammatory bowel disease
* Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
* Presence of uncontrolled infection
* Prolongation of corrected QT interval (QTc) > 480 msecs.
* History of any one of more of the following cardiovascular conditions within the past 6 months:
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Symptomatic peripheral vascular disease
* Class III or IV congestive heart failure as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg]. Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Blood pressure must be re-assessed on two occasions that are separated by a minimum of 24 hours. The mean SBP / DBP values from each blood pressure assessment must be < 140/90mmHg in order for a subject to be eligible for the study.
* History of cerebrovascular accident (CVA), pulmonary embolism or insufficiently treated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti coagulant agents (excluding therapeutic warfarin) for at least 6 weeks are eligible. As noted in Section 8.2, use of therapeutic levels of warfarin must have ended more than 14 days prior to first dose of study drug.
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding diathesis.
* Hemoptysis within 6 weeks prior to first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Is unable or unwilling to discontinue prohibited medications, as listed in Section 8.2, for 14 days or five half-lives (whichever is longer) of a drug prior to the first dose of study drug and for the duration of the study.
* Use of an investigational agent, including an investigational anti-cancer agent, within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug.
* Prior use of an investigational or licensed tyrosine kinase inhibitor that targets VEGF receptors. Note: Prior use of bevacizumab is allowed.
* Is now undergoing and/or has undergone in the 28 days immediately prior to first dose of study drug, any cancer therapy (surgery, tumor embolization, chemotherapy, radiation therapy, immunotherapy, biological therapy, or hormonal therapy). Note: For prior bevacizumab therapy, at least 40 days should have elapsed between last dose of bevacizumab and first dose of study drug.
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 (with the exception of Grade 2 alopecia) and/or that is progressing in severity.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib, erlotinib, or pemetrexed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-11-15 (Actual); Primary Completion 2009-09-04 (Actual); Study Completion 2009-09-04 (Actual)

PRIMARY OUTCOMES:
MTD regimen for each combination regimen in each arm of the study as determined by an evaluation of AEs and changes in laboratory values. The MTD = highest dosing regimen that results in dose limiting toxicity in <= 1 of 6 patients. | Through a minimum of two cycles of therapy for each subject

SECONDARY OUTCOMES:
Pharmacokinetic endpoints will be AUC, Cmax, tmax, and t1/2 of pazopanib, erlotinib, and pemetrexed and clearance of pemetrexed. | Through a minimum of two cycles of therapy for each subject
Tumor response using RECIST criteria. | Through a minimum of two cycles of therapy for each subject
Levels of circulating cytokine and angiogenic factors (CAF) biomarkers (such as IL-2, IL-10, VEGF, sVEGFR-2) in plasma will be determined.
Pharmacogenetics Endpoint: Genetic variants in candidate genes in the host DNA will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (3):
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Nashville, Tennessee
- GSK Investigational Site, Orbassano (TO), Piedmont, Italy

REFERENCES:
- [Background] Dy GK, Infante JR, Eckhardt SG, Novello S, Ma WW, Jones SF, Huff A, Wang Q, Suttle AB, Ottesen LH, Adjei AA, Burris HA 3rd. Phase Ib trial of the oral angiogenesis inhibitor pazopanib administered concurrently with erlotinib. Invest New Drugs. 2013 Aug;31(4):891-9. doi: 10.1007/s10637-012-9887-6. Epub 2012 Nov 8. PMID 23135778
- See also: Results for study VEG109607 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/VEG109607?search=study&study_ids=VEG109607#rs